CLINICAL TRIAL: NCT06813573
Title: Prospective Analysis of Circulating Nucleosomes in Patients Receiving a First Line Treatment for a Non-Hodgkin Lymphoma
Acronym: EVOLITION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A02716-39; 2023-3670 (Other: CSET number)
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Follicular Lymphoma; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving first line of treatment with a RCHOP 21 regimen (Experimental): All patients will receive first line of treatment with a RCHOP 21 regimen
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — A maximum of 4 tubes of 10ml will be collected: at baseline (before cycle 1), before each cycle (from 2 to 6 included), at the end of the treatment, and in case of relapse during follow-up period

SUMMARY:
The goal of this study is to prospectively follow the level of circulating nucleosomes in patients treated for a non-Hodgkin lymphoma and determine whether it correlates with the clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of diffuse large B cell lymphoma or follicular lymphoma, according to the WHO 2016 classification, requiring a first line of treatment with a RCHOP 21 regimen
* Agreement to participate after receiving oral and written information on the study

Exclusion Criteria:

* History of previous treatment for lymphoma (excluding localized low dose radiotherapy in the case of follicular lymphoma)
* Treatment with a chemotherapy regimen different from RCHOP21

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Prospective quantitative analysis of the level of circulating nucleosomes at baseline and during treatment in patients with diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL) | From enrollment to the end of the study (24 months of follow-up from beginning of treatment for each patient)

SECONDARY OUTCOMES:
Correlation between the level of circulating nucleosomes (number of cells) and the response to treatment as defined by international response criteria | From enrollment to the end of the treatment (6 cycles of 21 days)
  We would like to understand whether the more nucleosomes circulating, the more the patient responds to treatment.
Comparison between the results of molecular analysis of ctDNA and DNA extracted from nucleosomes | From enrollment to the end of the study (24 months of follow-up from beginning of treatment for each patient)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No